CLINICAL TRIAL: NCT04016168
Title: Idiopathic Pulmonary Fibrosis and Serum Bank
Acronym: FPI
Status: Completed | Type: Observational
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 35RC14_9722; 2014-A00268-39 (Other: Id-RCB)
Record Dates: First submitted 2019-07-08; First posted 2019-07-11 (Actual); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: Idiopathic Pulmonary Fibrosis; Lung Diseases, Interstitial
Keywords: Biomarkers; CD163
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis; Lung Diseases, Interstitial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — The aim of the study is to set up a biocollection of serum from patients in a context of idiopathic DILD
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with DILD: Patients will be recruited at the consultations of the Rennes Rare Lung Disease Competence Centre. These will be patients in stable condition or in acute exacerbation of IPF.
  Interventions: Biological: Blood sample collection

INTERVENTIONS:
Biological: Blood sample collection — Three additional blood tubes (3 x 8mL) will be collected for this study. They will be added to the traditional diagnostic assessment carried out for their IPF, during their consultation at the competence centre for rare lung diseases. These samples will be taken by a registered nurse in the presence and under the responsibility of the investigator.

SUMMARY:
Idiopathic pulmonary fibrosis (IPF) is the most common form of chronic idiopathic diffuse interstitial lung disease (DILD) in adults. It is a fibroproliferative, irreversible disease of unknown cause, usually progressive, occurring mainly from the age of 60 and limited to the lungs. IPF is a serious disease with a median survival rate at diagnosis of 3 years.

The aim of the study is to set up a biocollection of serum from patients in a context of idiopathic DILD and a possible or confirmed diagnosis of common interstitial lung disease by chest CT.

Patients will be recruited at the consultations of the Rennes Rare Lung Disease Competence Centre. These will be patients in stable condition or in acute exacerbation of IPF.

DETAILED DESCRIPTION:
This study will initially focus on circulating serum CD163 markers, but a broader proteomics approach could be considered in a second phase to look for other markers of lung diseases.

ELIGIBILITY:
Inclusion Criteria:

* Patients seen on an outpatient basis and in stable or acute condition
* Patient over 18 years of age.
* The inclusion criteria will be those edited by the American Thoracic Society (ATS) and the European Respiratory Society (ERS) to diagnosis IPF

Exclusion Criteria:

* Patients who are unable or unwilling to sign the consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be recruited at the consultations of the Rennes Rare Lung Disease Competence Centre. These will be patients in stable condition or in acute exacerbation of IPF.
Sampling Method: Non-Probability Sample
Enrollment: 903 (Actual)
Dates: Start 2014-10-22 (Actual); Primary Completion 2022-12-28 (Actual); Study Completion 2022-12-28 (Actual)

PRIMARY OUTCOMES:
Determination of circulating CD163 serum concentration | Through study completion, an average of 4 years
  Serum CD163 levels in patients with possible or certain DILD will be performed by ELISA technique (R&D Systems kit, Minneapolis, MN).

CONTACTS AND LOCATIONS:
Overall Officials: Stéphane JOUNEAU, MD, PhD, Principal Investigator — University Hospital of Rennes
Locations (1):
- Rennes University Hospital - Service de Pneumologie, Rennes, France

IPD SHARING:
Plan to Share IPD: No